CLINICAL TRIAL: NCT04064970
Title: Patient Acceptable Symptom State in Non-Surgical Management of Female Stress Urinary Incontinence
Brief Title: Patient Satisfaction Survey of Non-surgical Urinary Incontinence Treatment
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Erin Duecy, Professor, University of Rochester
Other Study IDs: RSRB72759
Record Dates: First submitted 2019-02-14; First posted 2019-08-22 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PASS Cohort
  Interventions: Behavioral: patient acceptable symptom state (PASS)

INTERVENTIONS:
Behavioral: patient acceptable symptom state (PASS) — The Severity Index for Urinary Incontinence, which documents incontinence frequency and severity, pelvic floor distress, patient global impression of severity and improvement, physical function, depression, sleep disturbance, anxiety, global health and ability to participate in social roles and activities.

SUMMARY:
The purpose of this study is to identify self-reported wellness following nonsurgical treatment of stress urinary incontinence. This will be done by correlating the response of "yes" on the patient acceptable symptom state (PASS) question to responses from other questionnaires regarding urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (> 18 years) seeking care for stress urinary incontinence at the URMC in Rochester, NY, DUMC in Durham, NC, Western New York (WNY) Urology Associates in Cheektowaga, NY, or at the UTMB in Galveston, TX.
* English-speaking
* Possess the ability to complete electronic patient reported outcome questionnaires and voiding diaries

Exclusion Criteria:

* Women who decline to participate in the study
* Women were unable to complete electronic patient reported outcome questionnaires
* Women with greater than stage II uterovaginal prolapse or post-hysterectomy prolapse.
* Women considered citizens of the European Union (EU), including EU citizens living in the United States.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be women over the age of 18 who desire nonsurgical management of stress urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
number of participants whose Urinary Distress Inventory-6 (UDI-6) score predict their Patient Acceptable Symptom State (PASS) answer | 6 weeks
  Each participant will be asked to complete the Urinary Distress Inventory 6 (UDI-6) after enrollment and again after 6 weeks. This is a short validated disease-specific patient reported outcome measuring urinary incontinence severity. The UDI-6 is a likert scale based questionnaire that calculates the mean of the scores and multiplies that mean by 25 to scale the instrument to an "actual score" with a range of 0 - 100. The higher the score the greater perceived negative impact on an individual's quality of life. The question "Considering all of the different ways that urinary leakage is affecting you, do you consider your current state to be satisfactory?" and provide a yes/no answer. Statistical analysis will then be performed to determine the threshold score at which one is likely to consider their symptoms to be acceptable, PASS "yes". Participants whose UDI score matches their PASS answer will be considered predicted and counted for this outcome measure.

SECONDARY OUTCOMES:
Mean Minimal important difference (MID) of the Urinary Distress Inventory 6 (UDI 6 ) as determined by the anchor-based method of analysis | baseline to 6 weeks
  The UDI-6 is a likert scale based questionnaire that calculates the mean of the scores and multiplies that mean by 25 to scale the instrument to an "actual score" with a range of 0 - 100 with a questions specifically related to stress urinary incontinence. The higher the score the greater perceived negative impact on an individual's quality of life The MID represents a clinically significant improvement in self-reported symptomatology. Anchor-based methods assess responsiveness in relation to an external event or rating to quantify the meaning of the particular degree of change. This is traditionally assessed by a moderate relationship noted using correlations between the negative score change and the external anchor. Participants will complete the UDI-6 at baseline and after 6 weeks. The MID will be defined by the mean score change reported by women who indicate improvement on the Patient Global Impression of severity (PGI-S) and Improvement (PGI-I).
Mean Minimal important difference (MID) of the Urinary Distress Inventory 6 (UDI 6 ) as determined by the distribution-bases method of analysis | 6 weeks
  The UDI-6 is a likert scale based questionnaire that calculates the mean of the scores and multiplies that mean by 25 to scale the instrument to an "actual score" with a range of 0 - 100 with a questions specifically related to stress urinary incontinence. The higher the score the greater perceived negative impact on an individual's quality of life The MID represents a clinically significant improvement in self-reported symptomatology. Distribution-based methods rely on the distribution of scores within a population and relate clinical significance to a change in magnitude at least equal to a statistical parameter of group data such as standard deviation (SD). This is traditionally assessed by including the effect size and standard error of measurement (SEM). A medium effect (0.5 SD) and a small effect size (0.2SD). The MID is estimated as 1 SEM.
Mean Minimal important difference (MID) of the Urinary Impact Questionnaire 7 (UIQ-7) as determined by the anchor-based method of analysis | baseline to 6 weeks
  The UIQ-7 is a likert scale based questionnaire that calculates the mean of the scores and multiplies that mean by 25 to scale the instrument to an "actual score" with a range of 0 - 100. The higher the score the greater perceived negative impact on an individual's quality of life. The MID represents a clinically significant improvement in self-reported symptomatology. Anchor-based methods assess responsiveness in relation to an external event or rating to quantify the meaning of the particular degree of change. This is traditionally assessed by a moderate relationship noted using correlations between the negative score change and the external anchor. Participants will complete the UDI-6 at baseline and after 6 weeks. The MID will defined by the mean score change reported by women who indicate improvement on the Patient Global Impression of severity (PGI-S) and Improvement (PGI-I).
Mean Minimal important difference (MID) of the Urinary Impact Questionnaire 7 (UIQ-7) as determined by the distribution-bases method of analysis | 6 weeks
  The UIQ-7 is a likert scale based questionnaire that calculates the mean of the scores and multiplies that mean by 25 to scale the instrument to an "actual score" with a range of 0 - 100. The higher the score the greater perceived negative impact on an individual's quality of life The MID represents a clinically significant improvement in self-reported symptomatology. Distribution-based methods rely on the distribution of scores within a population and relate clinical significance to a change in magnitude at least equal to a statistical parameter of group data such as standard deviation (SD). This is traditionally assessed by including the effect size and standard error of measurement (SEM). A medium effect (0.5 SD) and a small effect size (0.2SD). The MID is estimated as 1 SEM.

CONTACTS AND LOCATIONS:
Locations (1):
- University Urogynecology Associates, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided